CLINICAL TRIAL: NCT05500729
Title: Evaluation of Isometric Strength and Hamstring/Quadriceps Ratio in Healthy CrossFit Subjects
Brief Title: Hamstring/Quadriceps Ratio in CrossFit
Acronym: HQCROSS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Camila Velo Etcheverry (Other)
Responsible Party: Sponsor-Investigator, Camila Velo Etcheverry, PT Physiotherapy departament, Maimonides University
Organization: Maimonides University (Other)
Other Study IDs: 5738
Record Dates: First submitted 2022-08-08; First posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; Muscle Strength; Hamstring Muscles; Quadriceps Muscles; Young Adult; Isometric Contraction; Muscle Strength Dynamometer; Human physical conditioning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female CrossFitters: Crossfit practitioners born as female
  Interventions: Other: Hamstrings maximal voluntary isometric contraction.; Other: Quadriceps maximal voluntary isometric contraction
- Male CrossFitters: Crossfit practitioners born as male
  Interventions: Other: Hamstrings maximal voluntary isometric contraction.; Other: Quadriceps maximal voluntary isometric contraction

INTERVENTIONS:
Other: Hamstrings maximal voluntary isometric contraction. — Hamstrings maximal voluntary isometric contraction (MVIC) will be measured with an isometric dynamometer (3 reps x 5 sec work x 10 sec rest). The best rep will be used. Whenever the third one was the best, additional measurements will be taken until a decrease in torque will be obtained to determine the maximum.
Other: Quadriceps maximal voluntary isometric contraction — Quadriceps maximal voluntary isometric contraction (MVIC) will be measured with an isometric dynamometer (3 reps x 5 sec work x 10 sec rest). The best rep will be used. Whenever the third one was the best, additional measurements will be taken until a decrease in torque will be obtained to determine the maximum.

SUMMARY:
Crossfit® is a high-intensity physical training plan based on a program that includes exercises such as running, weight lifting and gymnastic movements. It focuses on the development of 10 physical qualities: strength, balance, cardiovascular and respiratory endurance, coordination, power, flexibility, agility, speed, precision and muscular endurance.Unfortunately, research on its effects is still at the beginning. The time of each session is one hour, which is divided into a warm-up of 10-30 minutes, strength training or skills, endurance work and finally a recovery phase, mobility and stretching. These types of exercises are incorporated into group training sessions called Workout of The Day (WOD).

Muscular strength is the action produced by a muscle or muscle group against resistance. It is one of the fundamental physical qualities for activities of daily living.

Digital isometric dynamometry is a tool to evaluate maximum voluntary isometric contraction (MVIC).

Hamstring muscles are responsible for hip extension and knee flexion. Moreover, they are the main protectors against anterior knee subluxation due to their action in conjunction with the anterior cruciate ligament (ACL).The quadriceps is one of the largest and most powerful muscles of the human body.

The ratio between hamstrings and quadriceps muscles has a strong correlation with lower limb injuries. This ratio, known as "H:Q" has proved to be the most reliable indicator to quantify a neuromuscular decompensation that causes an injury and, in addition, it is used as a prognostic indicator.

ELIGIBILITY:
Inclusion Criteria:

* Regular members of Tuluka Fitness Palermo.
* With at least 1 year of Crossfit training.

Exclusion Criteria:

* Subjects with a history of knee surgery.
* Who have any type of musculoskeletal injury to the dominant lower limb.
* Who suffer from neurological disorders.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of regular members of Tuluka Fitness Palermo, of both sex between 20 and 40 years of age, who have been training for more than 1 year on a recreational basis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-08-22 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Hamstrings maximal voluntary isometric contraction | Day 1
  Hamstrings force generated by the patient during a maximal voluntary isometric contraction, measured by an isometric dynamometer with load cell and computer interface.
  The best of the 3 repetitions will be considered. Whenever the third one is the best, additional measurements will be taken until a decrease in torque is obtained in order to determine the maximum.
  Unit: Newtons
Quadriceps maximal voluntary isometric contraction. | Day 1
  Quadriceps force generated by the patient during a maximal voluntary isometric contraction, measured by an isometric dynamometer with load cell and computer interface.
  The best of the 3 repetitions will be considered. Whenever the third one was the best, additional measurements will be taken until a decrease in torque is obtained in order to determine the maximum.
  Unit: Newtons

SECONDARY OUTCOMES:
Hamstring / Quadriceps Ratio | Day 1
  The ratio between hamstrings and quadriceps muscles has a strong correlation with lower limb injuries. This ratio, known as "H:Q" has proved to be the most reliable indicator to quantify a neuromuscular decompensation that causes an injury and, in addition, it is used as a prognostic indicator.
  Minimum value: -1 Maximum value: 1 A value below 0.6 indicates risk of injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Maimonides University, Buenos Aires, Buenos Aires F.D., Argentina